CLINICAL TRIAL: NCT01579058
Title: A Randomized Trial of Beta-blocker Therapy in Aortic Stenosis
Brief Title: Effect of Bisoprolol on Progression of Aortic Stenosis
Acronym: BLAST
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The sponsor discontinued to support the study.
Sponsor: Asan Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Duk-Hyun Kang, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-0884
Record Dates: First submitted 2012-04-14; First posted 2012-04-17 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Aortic Stenosis
Keywords: aortic stenosis; beta-blocker
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Bisoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bisoprolol (Active Comparator): bisoprolol 5mg qd
  Interventions: Drug: bisoprolol
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: bisoprolol — bisoprolol 5mg qd for 4 years
  Other Names: Concor
  Arms: bisoprolol
Drug: placebo — placebo for 4 years
  Arms: placebo

SUMMARY:
Aortic stenosis has been thought to be a degenerative process basically induced by long-lasting mechanical stress, and hemodynamic factors such as shear forces, acceleration of blood flow, hypertension and rapid heart rate might contribute to progression of aortic stenosis. Peak aortic jet velocity is known to be associated with clinical outcomes in mild and moderate AS, and our previous study showed that rate of progression was significantly associated with baseline aortic jet velocity in mild aortic stenosis. Because beta-blocker therapy would decrease aortic jet velocity and heart rate, it might decrease hemodynamic stress and eventually slow down the degenerative process in patients whose disease is not too advanced for therapy to be effective. The investigators hypothesized that a beta-blocker therapy would decrease the rate of progression of aortic stenosis by modifying hemodynamic factors favorably in patients with mild to moderate aortic stenosis.

DETAILED DESCRIPTION:
Aortic stenosis (AS) is a gradually progressive disease, characterized by an increase in calcium deposition leading to progressive narrowing of the aortic valve (AV). There are currently no effective medical treatment to halt the disease process and surgical valve replacement remains the only proven therapy when the valve becomes severely stenotic. AS is mediated by a chronic inflammatory disease process, very similar to that seen in atherosclerosis, but lipid-lowering therapy did not slow the progression of AS in the SALTIRE, SEAS, or ASTRONOMER trials. It is possible that these trials may have targeted patients in whom disease was too advanced for lipid-lowering therapy to be effective, or in whom atherosclerotic mechanism was not the central pathogenic process in AS. Because identifying and treating patients in earlier stages of AS would not be cost-effective, it seems more logical to explore alternative pharmacological approaches.

AS has been thought to be a degenerative process basically induced by long-lasting mechanical stress, and hemodynamic factors such as shear forces, acceleration of blood flow, hypertension and rapid heart rate might contribute to progression of AS. Peak aortic jet velocity is known to be associated with clinical outcomes in mild and moderate AS, and our previous study showed that rate of progression was significantly associated with baseline aortic jet velocity in mild AS. Because beta-blocker therapy would decrease aortic jet velocity and heart rate, it might decrease hemodynamic stress and eventually slow down the degenerative process in patients whose disease is not too advanced for therapy to be effective. In a retrospective, observational study, beta-blocker therapy was associated with a favorable clinical outcome in AS.

The investigators hypothesized that bisoprolol, a new generation beta-blocker, would decrease the rate of progression of AS by modifying hemodynamic factors favorably in patients with mild to moderate AS.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate aortic stenosis defined by peak velocity of aortic jet between 2.0 and 3.5 m/sec
* Untreated hypertension: systolic BP ≥ 140 or diastolic BP ≥ 90 mmHg Treated hypertension using dihydropiridine calcium channel blockers, ACE inhibitors, ARB or diuretics
* Patients received no beta-blocker therapy for more than 12 months

Exclusion Criteria:

* Symtomatic aortic stenosis: presence of exertional dyspnea, angina or syncope
* Planned cardiac surgery (e.g., CABG, valve repair or replacement, or aneurysmectomy) or planned major non-cardiac surgery within the study period
* Stroke or resuscitated sudden death in the past 6 months
* Evidence of congestive heart failure, or left ventricular ejection fraction < 50%
* Significant renal disease manifested by serum creatinine > 2.0mg/dL
* History of intolerance to beta-blocker
* History of adult asthma manifested by bronchospasm in the past 6 months, or currently taking regular anti-asthmatic medication(s)
* Moderate or severe aortic regurgitation
* Atrial fibrillation
* Female of child-bearing potential who do not use adequate contraception and women who are pregnant or breast-feeding
* A diagnosis of cancer (other than superficial squamous or basal cell skin cancer) in the past 3 years or current treatment for the active cancer
* Any clinically significant abnormality identified at the screening visit, physical examination, laboratory tests, or electrocardiogram which, in the judgment of the Investigator, would preclude safe completion of the study
* Unwillingness or inability to comply with the procedures described in this protocol

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in peak aortic jet velocity from baseline to 4 years follow-up | 4 years
  Change in peak aortic jet velocity from baseline to 4 years follow-up. For each patient, the change in peak aortic jet velocity is calculated as (peak aortic jet velocity at 4 year follow-up) - (peak aortic jet velocity at baseline) on Doppler echocardiography.

SECONDARY OUTCOMES:
Change in mean pressure gradient across aortic valve | 4 years
  Change in mean pressure gradient across aortic valve from baseline to 4 years follow-up
Change in aortic valve area | 4 years
  Change in aortic valve area from baseline to 4 years follow-up
Change in BNP levels | 4 years
  Change in BNP levels from baseline to 4 years follow-up
Change in E/E' ratio | 4 years
  Change in the ratio of E velocity (early mitral inflow velocity) to E' velocity (early mitral annular velocity) from baseline to 4 years follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Duk-Hyun Kang, M.D., Principal Investigator — Asan Medical Center
Locations (3):
- South Korea (3):
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul